CLINICAL TRIAL: NCT06368986
Title: An Open Label, Phase 1 Study to Assess the Effect of Food on Bioavailability for an Investigational Capsid Inhibitor in Healthy Adult Participants
Brief Title: A Study to Investigate the Effect of Food on the Bioavailability of a Capsid Inhibitor (CAI) in Male and Female Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 222420
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: HIV Infections
Keywords: Fasted condition; Fed condition; Bioavailability; Capsid inhibitor; VH4011499
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part 1 Dose A - Fasted condition (Experimental): VH4011499 Dose A tablet administered in fasted condition.
  Interventions: Drug: VH4011499 Dose A
- Part 1 Dose A- Fed condition (high fat meal) (Experimental): VH4011499 Dose A tablet administered in fed condition (high fat meal).
  Interventions: Drug: VH4011499 Dose A
- Part 2 Dose B - Optional - Fed condition (low fat meal) (Experimental): VH4011499 Dose B tablet administered in fed condition (low fat meal).
  Interventions: Drug: VH4011499 Dose B
- Part 3 Dose B - Fasted condition (Experimental): VH4011499 Dose B tablet administered in fasted condition.
  Interventions: Drug: VH4011499 Dose B
- Part 3 Dose B - Fed condition (high fat meal) (Experimental): VH4011499 Dose B tablet administered in fed condition (high fat meal).
  Interventions: Drug: VH4011499 Dose B

INTERVENTIONS:
Drug: VH4011499 Dose A — VH4011499 administered in fasted or fed conditions.
  Arms: Part 1 Dose A - Fasted condition; Part 1 Dose A- Fed condition (high fat meal)
Drug: VH4011499 Dose B — VH4011499 Dose B administered in fasted or fed conditions.
  Arms: Part 2 Dose B - Optional - Fed condition (low fat meal); Part 3 Dose B - Fasted condition; Part 3 Dose B - Fed condition (high fat meal)

SUMMARY:
The purpose of this study is to evaluate effect of food (in fasted and fed conditions) on the bioavailability of CAI VH4011499.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are 18 to 55 years of age.
* Participants who are overtly healthy.
* One SARs-CoV-2 negative test is required prior to dosing
* Body weight within 50-100 kg and body mass index (BMI) within the range 19-32 kg/m2 (inclusive).
* Capable of giving signed informed consent.
* Participants male at birth must use male condoms, and participants female at birth who are of childbearing potential must be using acceptable forms of birth control.

Exclusion Criteria:

* History or presence of disorders capable of significantly altering the absorption, metabolism, or elimination of drugs.
* Current or chronic liver disease, hepatic or biliary abnormalities, or relevant hepatitis.
* Abnormal blood pressure.
* Any malignancy within the past 5 years except certain localized malignancies, or breast cancer within the past 10 years. Participants with exclusionary electrocardiogram findings.Positive HIV test or ongoing behaviors that put the participant at high risk for HIV acquisition.
* Participants who are breastfeeding or plan to become pregnant during the study.
* Past or intended use of exclusionary medications or vaccines.
* Exposure to >4 new investigational products within 12 months, previous participation in this study, or current enrolment or participation in another investigational study.
* ALT >1.5x upper limit of normal (ULN), total bilirubin >1.5x ULN, and/or estimated serum creatinine clearance <60 mL/min.
* History of or current infection with hepatitis B or hepatitis C.
* Positive SARS-CoV-2 test, having signs and symptoms suggestive of COVID-19, or contact with known COVID-19 positive person.
* Positive HIV antibody test.
* Participants with positive results for illicit drug use, regular use of drugs of abuse, tobacco or nicotine-containing product use, and/or excessive alcohol use.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration - time curve from time zero (pre-dose) to infinity time (AUC[0-inf]) of VH4011499 | From Day 1 (pre-dose) to Day 28
Area under the plasma drug concentration - time curve from zero (pre-dose) to the end of the dosing interval at steady state (AUC[0-tlast) of VH4011499 | From Day 1 (pre-dose) to Day 28
Maximum observed plasma drug concentration (Cmax) of VH4011499 | From Day 1 (pre-dose) to Day 28
Time to maximum observed plasma concentration (Tmax) of VH4011499 | From Day 1 (pre-dose) to Day 28

SECONDARY OUTCOMES:
Number of participants with AEs (Adverse Events), by severity | From Day 1 (pre-dose) to Day 28
  An AE is any untoward medical occurrence in a participant or clinical investigation participant and can be any sign, symptom, or disease temporally associated with the use of a medicinal product. The severity scale is assessed as following: Grade 1 = mild symptoms causing no or minimal interference with usual social and functional activities with intervention not indicated. Grade 2 = moderate symptoms causing greater than minimal interference with usual social and functional activities with intervention indicated. Grade 3 = severe symptoms causing inability to perform usual social and functional activities with intervention or hospitalization indicated. Grade 4 = potentially life-threatening symptoms causing inability to perform self-care functions with intervention indicated to prevent permanent impairment, persistent disability, or death, Grade 5 = death.
Number of participants with maximum toxicity grade increase from baseline for liver laboratory parameters | From Day 1 (pre-dose) to Day 28
  The assessed laboratory assessments include Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), alkaline phosphatase (ALP), direct bilirubin and total bilirubin, in both fed and fasted conditions.
Change from baseline in liver panel parameters: total bilirubin and direct bilirubin (micromoles per liter) | From Day 1 (pre-dose) to Day 28
Change from baseline in liver panel parameters: ALT, ALP and AST (International units per liter) | From Day 1 (pre-dose) to Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf